CLINICAL TRIAL: NCT05195892
Title: A Single-center, Randomized, Open-label, Three-period Crossover Study to Investigate the Bioequivalence of Alpelisib Granule and Film-coated Tablet Formulation, and the Food Effect of Alpelisib Granule Formulation in Adult Healthy Volunteers
Brief Title: Investigate Bioequivalence of Alpelisib Granule and Film-coated Tablet Formulation and the Food Effect of Alpelisib Granule Formulation in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719F12101
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers
Keywords: adult; bioequivalence; food effect; three-period six sequence crossover; alpelisib; BYL719

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive a single oral dose of alpelisib film-coated tablet at 50 mg in fed state (treatment A) in period 1 followed by a single oral dose of alpelisib granule at 50 mg in fed state (treatment B) in period 2 and a single oral dose of alpelisib granule at 50 mg in fasted state (treatment C) in period 3.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 2 (Experimental): Participants will receive a single oral dose of alpelisib granule at 50 mg in fed state (treatment B) in period 1 followed by a single oral dose of alpelisib granule at 50 mg in fasted state (treatment C) in period 2 followed by a single oral dose of alpelisib film-coated tablet at 50 mg in fed state (treatment A) in period 3.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 3 (Experimental): Participants will receive a single oral dose of alpelisib granule at 50 mg in fasted state (treatment C) in period 1 followed by a single oral dose of alpelisib film-coated tablet at 50 mg in fed state (treatment A) in period 2 followed by a single oral dose of alpelisib granule at 50 mg in fed state (treatment B) in period 3.
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 4 (Experimental): Participants will receive a single oral dose of alpelisib granule at 50 mg in fasted state (treatment C) in period 1 followed by a single oral dose of alpelisib granule at 50 mg in fed state (treatment B) in period 2 followed by a single oral dose of alpelisib film-coated tablet at 50 mg in fed state (treatment A).
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 5 (Experimental): Participants will receive a single oral dose of alpelisib film-coated tablet at 50 mg in fed state (treatment A) in period 1 followed by a single oral dose of alpelisib granule at 50 mg in fasted state (treatment C) in period 2 followed by a single oral dose of alpelisib granule at 50 mg in fed state (treatment B).
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 6 (Experimental): Participants will receive a single oral dose of alpelisib granule at 50 mg in fed state (treatment B) in period 1 followed by a single oral dose of alpelisib film-coated tablet at 50 mg in fed state (treatment A) in period 2 followed by a single oral dose of alpelisib granule at 50 mg in fasted state (treatment C).
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — Single oral dose of alpelisib film-coated tablet at 50 mg in fed state
Drug: Treatment B — Single oral dose of alpelisib granule at 50 mg in fed state
Drug: Treatment C — Single oral dose of alpelisib granule at 50 mg in fasted state

SUMMARY:
The purpose of this study is to assess bioequivalence of the granule formulation of alpelisib as compared to the film-coated tablet formulation in healthy volunteers in the fed state. In addition, the food effect of the granule formulation will be investigated between the fed state and the fasted state.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, three-period six-sequence crossover study.

The study consists of a screening period followed by Periods 1, 2, and 3 and a safety follow-up. Randomization occurs at the beginning of Period 1, whereby every participant who passes the screening will be randomized to one of 6 sequences with 1:1:1:1:1:1 randomization ratio. Each sequence consists of a permutation of three treatments: A, B and C. The order of the sequence of the treatments (A, B, C) will be determined by randomization to the assigned sequence.

A total of 60 participants will be enrolled with approximately 10 participants per sequence, in order to obtain at least 48 evaluable participants for comparison of the granule formulation in fed status and the film-coated tablet formulation in fed status.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 and 55 years of age
* Female participants must be postmenopausal or not of child bearing potential.
* Participants must weigh 50 kg - 120 kg and have BMI= 18.0-30.0 kg/m2
* Participants should be in good health as determined by no clinically significant findings from the medical history, physical examination, vital signs, and ECG.
* Participant must have laboratory values (including fasting plasma glucose and HgbA1C) within the reference range at the local laboratory
* At screening, and at baseline visit of each Period, participant has vital signs which are within the protocol defined ranges

Exclusion Criteria:

* Women of childbearing potential
* Sexually active male participant with partner(s) of women of childbearing potential, UNLESS agree to comply with highly effective contraception AND use a condom
* Participant with
* significant illness, including infections, or hospitalization within the 30 days prior to dosing.
* diabetes mellitus or participants with fasting plasma glucose (FPG) levels > 100 mg/dL or >5.55 mmol/L.
* clinically significant risk of developing diabetes mellitus during the study
* Use of:
* tobacco products within 3 months prior to first dosing
* drug or alcohol abuse within 12 months prior to first dose
* alcohol within 48 hours prior to the dosing of each treatment period.
* any prescription or non-prescription, herbal medication, dietary supplements or vitamins during 14 days prior to dosing..
* History of :
* clinically significant hematologic, renal, endocrinologic, pulmonary, cardiovascular, hepatic, or allergic disease, medically documented. including uncontrolled hypertension, interstitial lung disease, or other causes of dyspnea, acute pancreatitis within 1 year of screening or past medical
* chronic pancreatitis.
* cardiac disease
* immunodeficiency diseases
* malignancy of any organ system carcinoma of the skin or in situ cervical cancer), within 5 years,
* erythema multiform (EM), Steven-Johnson-Syndrome (SJS) or Toxic Epidermal Necrolysis (TEN).
* history or presence of
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs.
* clinically significant ECG abnormalities or a family prolonged QT-interval syndrome.
* chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV).

Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of alpelisib for Treatment A and Treatment B | Period 1, 2 and 3 at pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12. 24, 48, 72 and 96 hours post-dose
  Blood samples will be collected at specified time points to compare Cmax of the test formulation (Treatment B: granule formulation in fed state) versus the reference formulation (Treatment A: the film-coated tablet formulation in fed state). PK parameters will be calculated using noncompartmental data analysis of plasma concentration-time data

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of alpelisib for Treatment B and Treatment C | Period 1, 2 and 3 at pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12. 24, 48, 72 and 96 hours post-dose
  Blood samples will be collected at specified time points to compare Cmax of the granule formulation in the fed state (Treatment B) versus the granule formulation in the fasted state (Treatment C). PK parameters will be calculated using noncompartmental data analysis of plasma concentration-time data.
Area under plasma concentration time curve (AUC) from zero to 96 hours post dose of alpelisib for Treatment A, Treatment B and Treatment C | Period 1, 2 and 3 at pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12. 24, 48, 72 and 96 hours post-dose
  Blood samples will be collected at specified time points to calculate AUC0-96 of alpelisib after a single oral dose of alpelisib film coated tablet formulation in fed state (Treatment A), after a single oral dose of alpelisib granule formulation in fed state (Treatment B), after a single oral dose of alpelisib granule formulation in fasted state (Treatment C). PK parameters will be calculated using noncompartmental data analysis of plasma concentration-time data

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burmeister Getz E, Niglis S, Papadimitriou A, Statelova M, Ren X, Nakhla K, Sharaby S, Tariq M, Garbuio L, Bakhsh S. Predicting and Confirming Bioequivalence of Alpelisib Oral Granules and Tablets for Patients With PIK3CA-Related Disorders. AAPS PharmSciTech. 2025 Apr 30;26(5):121. doi: 10.1208/s12249-025-03109-4. PMID 40307580